CLINICAL TRIAL: NCT06433999
Title: A 12-Week Open-Label Pilot Study to Investigate the Efficacy and Safety of Oral Brepocitinib in Adults With Skin-Predominant Dermatomyositis
Brief Title: A 12-Week Open-Label Study to Investigate the Efficacy and Safety of Brepocitinib in Adults With Skin-Predominant Dermatomyositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Priovant Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVT-2201-202
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Dermatomyositis; Dermatomyositis, Adult Type
Keywords: skin-predominant dermatomyositis; dermatomyositis
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brepocitinib (Experimental)
  Interventions: Drug: Brepocitinib

INTERVENTIONS:
Drug: Brepocitinib — Oral Brepocitinib PO QD

SUMMARY:
This is a prospective, 12-week, open-label, single-arm study. The study population comprises individuals with refractory skin disease characteristic of dermatomyositis with no to minimal muscle involvement. After an up to 8-week Screening Period, eligible participants will receive brepocitinib 30 mg orally (PO) QD for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of dermatomyositis according to 2017 EULAR/ACR Classification Criteria for Idiopathic Inflammatory Myopathies
* Active cutaneous manifestations of dermatomyositis
* Adult subjects (18-75 years old)
* Weight > 40 kg to < 130 kg, and with a body mass index (BMI) < 40 kg/m2.

Exclusion Criteria:

* Dermatomyositis with end-stage organ involvement
* Dermatomyositis with irreversible muscle involvement

History of:

* Any lymphoproliferative disorder
* Active malignancy;
* History of cancer within 5 years prior to randomization (exceptions for basal cell carcinoma, squamous cell carcinoma, ductal carcinoma in situ of the breast, carcinoma in situ of the uterine cervix, or thyroid carcinoma.) Cancer-associated dermatomyositis
* Overlap myositis/connective tissue disease (except for overlap with Sjögren's syndrome)
* Participants at a risk of thrombosis or cardiovascular disease
* Participants with a high risk for herpes zoster reactivation
* Participants with active or recent infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in CDASI-A score from baseline through Week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mangold, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Clinical Trial Site, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No